CLINICAL TRIAL: NCT00356382
Title: Decreasing Rates of Illnesses in Kids (DRINK)
Brief Title: Decreasing Rates of Illness in Kids (DRINK)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Dannon Company, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2006-291
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2007-04

CONDITIONS: Healthy
Keywords: probiotic; Lactobacillus (L.) casei; cultured dairy drink; Health
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lactobacillus (L.) casei

SUMMARY:
The purpose of this study is to determine the effectiveness of a cultured dairy drink with high concentrations of active L casei to reduce the cumulative rate of illness in daycare/school children ages 3 to 6.

DETAILED DESCRIPTION:
Probiotics are live microorganisms, which when administered in sufficient amounts, may improve health. Often, probiotics are ingested as supplements in powder, pill, or liquid form, designed specifically for medicinal benefit. Such supplements used in children have shown some potential benefits in the treatment and prevention of various diseases, including diarrhea, asthma, necrotizing enterocolitis and allergies.

In the past few years, interest has increased in the health-enhancing role f specific foods, referred to as functional foods- foods providing health benefits beyond their nutritional value. Yogurt, a fermented milk product produced by the action of two bacteria, Lactobacillus (L.) bulgaricus and Streptococcus (S.) thermophilus, is a functional food. In fact, two-thirds of primary care physicians, who counsel patients about nutrition, recommend consuming yogurt containing live active cultures for their patients' health benefit. However, evidence for these health outcomes is not sufficiently strong.

Daycare and school centers are ideal places for the transmission of respiratory infections and childhood diarrhea, often resulting in many missed days of both daycare and parental work. Illnesses related to daycare centers have been estimated to cost $1.8 billion per year in the United States. One of the primary purposes of daycare is to allow parents to work while their child is taken care of, thus, absences due to illnesses have many direct and indirect associated costs. Unfortunately, children in daycare centers have been shown to have more outpatient doctor visits, emergency room visits, and increased usage of prescription medicines than children in daycare.

Our overall goal is to study a cultured dairy drik with an efficacious probiotic at doses that result in probiotic survival in the gastrointestinal tract and subsequently reduce illnesses in daycare/school children ages 3-6.

The rationale for focusing on a drink as a vehicle for transmission of probiotics, is that it has the potential for a much greater public health impact than using probiotics in a medicinal manner, such as pills or capsules. Yogurt and yogurt like probiotic drinks are well established and popular with children and parents, a product that traditionally provides live cultures to the diet, and can provide protein, vitamins and minerals that are nutritious for the child. Additionally, these drinks are relatively inexpensive, widely available, and easy to ingest even for individuals with lactose intolerance. These positive attributes make it an idea carrier to deliver the health benefits of probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 3 to 6 years
* Attending daycare centers or school 5 days a week
* Subjects or parents/legal guardians who agree to have their child refrain from consuming dairy fermented products during the course of the study

Exclusion Criteria:

* Subjects whose caregivers do not speak English or Spanish
* Subjects with allergy or hypersensitivity to milk proteins or dairy food components like lactose
* Subjects that do not have proper storage facility for product to be held at home
* Subjects presenting with a chronic disease that requires daily medication (Ex. cancer, tuberculosis, Crohns disease, cirrhosis, multiple sclerosis, Type 1 Diabetes...)
* Subjects with cardiac, respiratory, or renal insufficiencies
* Subjects with chronic immunodeficiency (ex: HIV, Chemotherapy...)
* Subjects presenting any infection in the last 7 days
* Subjects with any current or past severe gastrointestinal or metabolic disease (malabsorption, ulcer, celiac disease...)
* Subjects with a history of severe respiratory disease that requires daily usage of medicine
* Subjects that used laxatives in the last 7 days
* Subjects currently with diarrhea or constipation in the last 7 days
* Subjects under artificial nutrition or that were under artificial nutrition in the last 2 months
* Subjects with special medicated diet (obesity, anorexia, metabolic pathology...)
* Subjects with eating disorders (anorexia, bulimia...)
* Subjects currently receiving, or that received in the last 7 days, any antibiotics, antiseptics, antifungals, corticosteroids, vaccines, anti histamines, non steroid anti-inflammatory drugs
* Subjects that had a gastro-intestinal surgery in the last 3 months
* Subjects that had any surgery or intervention requiring general anaesthesia in the last month
* Subjects enrolled in another clinical study, currently or during the last 2 months (exclusion period from the former study)
* Subjects presenting congenital malformation
* Subjects with failure to thrive, growth retardation, or any developmental problem
* Subjects not attending day care centers or schools 5 days a week
* Subjects who cannot obtain both of their parents/legal guardians' signatures if they are separated/divorced and have joint custody of the child

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 638
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Mean of sick days due to upper-respiratory and gastro-intestinal infections and diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Merenstein, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Department of Family Medicine, Washington D.C., District of Columbia, United States